CLINICAL TRIAL: NCT01577290
Title: An Internet-administered, Mindfulness Training Program for the Treatment of Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Per Carlbring, PhD, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMA
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Anxiety; Depression; Insomnia
Keywords: Anxiety; Depression; Insomnia; Mindfulness; Internet
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness training (Experimental): Group receives mindfulness training.
  Interventions: Behavioral: Internet-administered Mindfulness Training Program
- Discussion group (Active Comparator): Group has access to a discussion group.
  Interventions: Behavioral: Discussion group

INTERVENTIONS:
Behavioral: Internet-administered Mindfulness Training Program — A 10 week, internet-administered mindfulness training program, featuring no therapist-support. 10 minutes of training, twice per day.
  Arms: Mindfulness training
Behavioral: Discussion group — Access to a discussion group with the possibility of sharing experiences, methods of relief, and the like.
  Arms: Discussion group

SUMMARY:
The purpose of this study is to examine the effects of a 10 week mindfulness training program -- without therapist-support -- as treatment of anxiety. Effects on depression, quality of life, and insomnia symptoms will also be studied.

DETAILED DESCRIPTION:
Previous research has provided evidence for the thesis that training in mindfulness can decrease symptoms of anxiety and depression. This study will examine the effects of a 10 week mindfulness training program -- without therapist-support -- as treatment of anxiety. Effects on depression, quality of life, and insomnia symptoms will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy DSM-IV criteria for an anxiety disorder
* Living in Sweden and being able to read Swedish
* Access to computer with internet connection

Exclusion Criteria:

* Currently receiving other psychological treatment
* Non-stable use of psychoactive medication
* Deemed suicidal
* Deemed to suffer from other psychological disorder, e.g. psychosis, bipolarity etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Beck Anxiety Inventory (BAI) | 24 hours
  21 item rating scale for anxiety symptoms.
Change from baseline in Beck Anxiety Inventory (BAI) | 6 months
  21 item rating scale for anxiety symptoms.

SECONDARY OUTCOMES:
Change from baseline in Beck Depression Inventory (BDI) | 24 hours
  21 item rating scale for depression symptoms.
Change from baseline in Beck Depression Inventory (BDI) | 6 months
  21 item rating scale for depression symptoms.
Change from baseline in Quality Of Life Inventory (QOLI) | 24 hours
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 6 months
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Insomnia Severity Index (ISI) | 24 hours
  7 item rating scale of insomnia symptoms.
Change from baseline in Insomnia Severity Index (ISI) | 6 months
  7 item rating scale of insomnia symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, Professor, Principal Investigator — Department of Psychology, Umeå University
Locations (1):
- Department of Psychology, Umeå University, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Result] Boettcher J, Astrom V, Pahlsson D, Schenstrom O, Andersson G, Carlbring P. Internet-based mindfulness treatment for anxiety disorders: a randomized controlled trial. Behav Ther. 2014 Mar;45(2):241-53. doi: 10.1016/j.beth.2013.11.003. Epub 2013 Nov 25. PMID 24491199